CLINICAL TRIAL: NCT02000882
Title: Phase II Multicenter Single-arm Study of BKM120 Plus Capecitabine for Breast Cancer Patients With Brain Metastases
Brief Title: STAR Cape+BKM120 MBC With Brain Met
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Oncology Research (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11025; CBKM120ZUS39T (Other: Novartis)
Record Dates: First submitted 2013-11-26; First posted 2013-12-04 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Brain Metastases; Breast Cancer; Metastatic Breast Cancer
Keywords: Breast Cancer; Triple Negative Breast Cancer; Brain Metastases; Capecitabine; Metastatic Breast Cancer
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — NVP-BKM120; Capecitabine; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BKM120 plus Capecitabine (Experimental): BKM120 will be administered at a dose of 100 mg orally (PO) daily. Capecitabine will be administered at a dose of 1000 mg/m2 orally (PO) twice a day (rounded down to the nearest 500 mg pill) 14 days on and 7 days off.
  For patients with HER2+ MBC only, standard every 3-weekly trastuzumab (6 mg/kg IV) will be added to the capecitabine/BKM120.
  Interventions: Drug: BKM120; Drug: capecitabine; Drug: Trastuzumab

INTERVENTIONS:
Drug: BKM120
  Other Names: buparlisib
Drug: capecitabine
  Other Names: Xeloda
Drug: Trastuzumab
  Other Names: Herceptin

SUMMARY:
This is a study to determine the safety and effectiveness of BKM120 plus capecitabine in breast cancer patients with brain metastases.

Both capecitabine and BMK120 have previously shown activity in patients with breast cancer. Like capecitabine, BMK120 is also effective in crossing the blood brain barrier making it a preferred candidate for its evaluation in patients with metastatic breast cancer (MBC).

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, single-arm study to determine the safety and efficacy of BKM120 plus capecitabine in breast cancer patients with brain metastases. 40 patients will be included, who have either ER+/HER2-, HER2+ or triple negative breast cancer..

The Graded Prognostic Assessment (GPA) is a recently developed, validated prognostic score for patients with brain metastases. The Graded Prognostic Assessment will be utilized to evaluate efficacy in this clinical study.

Capecitabine is a prodrug which is enzymatically converted to 5-fluorouracil in its tumor target where it inhibits DNA synthesis and slows tumor growth. It is currently FDA approved for both colorectal and breast cancer. BMK120 is a pan phosphatidylinositol-3-kinase inhibitor being developed under IND# 102,823 by Novartis Corporation. As of September 2012 over 600 patients had been enrolled in fourteen separate Novartis sponsored monotherapy or combination therapy clinical studies of BMK120.

Phosphatidylinositol-3-kinase (PI3K) signaling regulates diverse cellular functions including cell proliferation, survival, translational regulation of protein synthesis, glucose metabolism, cell migration, and angiogenesis. PI3K signaling also serves a central role in the pathogenesis of numerous cancers.

Constitutive activation of PI3K signaling is known to be a critical step in mediating the transforming potential of oncogenes and tumor suppressors in many tumor types. Resistance to a variety of therapeutic interventions, including hormonal therapy, anti-HER2 therapies and chemotherapy can also be linked to constitutive activation of the PI3K pathway.

Preliminary data suggest that activation of the PI3K pathway is a predictor of a poor prognostic outcome in many cancer types. Thus, as a pan-PI3K inhibitor, BMK120 may provide a therapeutic benefit to patients with MBC. Both capecitabine and BMK120 have previously shown activity in patients with MBC. Like capecitabine, BMK120 is also effective in crossing the blood brain barrier making it a preferred candidate for its evaluation in patients with MBC.

Trastuzumab is a monoclonal antibody that targets the HER2 receptor which is overexpressed or amplified in approximately 20-25% of breast cancers. The clinical benefit of trastuzumab in women with metastatic breast cancer has been demonstrated in two pivotal studies.

Current clinical experience with BMK120 has shown that its most frequent adverse events (AEs) include fatigue, decreased appetite, diarrhea, hyperglycemia, nausea, rash and mood alteration disorders. Therefore patients will be closely monitored for fasting plasma glucose (FPG) HbA1c, and insulin C-peptide. Patients will also be frequently and routinely evaluated for mood disorders and disturbances. The remaining most frequent AEs will be detected by regular, frequent monitoring with symptomatic treatment to be provided as required.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Female
3. Histologically and/or cytologically confirmed diagnosis of inoperable metastatic breast cancer
4. ER+/HER2- OR HER2+ OR triple-negative breast cancer, assessed as ER-, PgR-, and HER2-negative by local laboratory testing; HER2 negative status (based on most recently analyzed biopsy) is defined as IHC status of 0, 1+ or 2+ (if IHC 2+, a negative FISH test is required, ie, HER2 FISH ratio < 2.0); ER-negative and PR-negative status is defined as ER and PgR <10% nuclei positive by IHC. HER2-positive status is defined as 3+ staining in ≥10% of cells by immunohistochemistry or a HER2/CEP17 ratio ≥2 or an average of ≥6 HER2 gene copies per cell by in situ hybridization (ISH)
5. At least one CNS lesion that is at least 5mm in size in at least one dimension in the setting of prior WBRT

   * Prior WBRT is required and may have been administered at any time in patient's treatment history. Patients in the primary analysis will not have evidence of progression of disease following WBRT. However, patients whose brain metastases have progressed following WBRT are eligible. Patients must have completed WBRT at least 3 weeks prior to study entry.
   * Prior SRS is allowed, but previous treatment of the 5mm target CNS lesion with SRS is not permitted
6. ECOG performance status ≤ 2
7. Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hb >9 g/dL
8. Total calcium (corrected for serum albumin) within normal limits (biphosphonate use for malignant hypercalcemia control is not allowed)
9. Magnesium ≥ the lower limit of normal
10. Potassium within normal limits for the institution
11. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within normal range (or ≤ 3.0 x upper limit of normal (ULN) if liver metastases are present)
12. Serum bilirubin within normal range (or ≤ 1.5 x ULN if liver metastases are present; or total bilirubin ≤ 3.0 x ULN with direct bilirubin within normal range in patients with known Gilbert Syndrome)
13. Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
14. Serum amylase ≤ ULN
15. Serum lipase ≤ ULN
16. Fasting plasma glucose ≤ 120 mg/dL (6.7 mmol/L)
17. Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
18. INR ≤ 2
19. Life expectancy > 12 weeks
20. Available tissue (blocks and/or slides) samples unless discussed in advance with study principal investigator
21. Patient is able to swallow and retain oral medication
22. Signed most recent patient informed consent form
23. Signed Patient Authorization Form

Exclusion Criteria:

1. Patient received prior treatment with a P13K inhibitor.
2. Patient with known hypersensitivity to BKM120, capecitabine, or their excipients.
3. Patient has evidence of impending herniation on baseline brain imaging.
4. Patient has evidence of diffuse leptomeningeal disease on brain MRI or by previously documented CSF.
5. Patient has acute or chronic liver, renal disease or pancreatitis (liver metastases are allowed)
6. Patients has a mood disorder as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire (PHQ-9 and/or GAD-7):

   * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others) or patients with active severe personality disorders (defined according to DSM- IV) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug.
   * ≥ CTCAE grade 3 anxiety
   * Meets the cut-off score of ≥ 12 in the PHQ-9 or a cut-off of ≥ 15 in the GAD-7 mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
7. Patients has diarrhea ≥ CTCAE grade 2
8. Patients with uncontrolled hypertension defined as systolic blood pressure 170 or greater or diastolic blood pressure over 100.
9. Patient has active cardiac disease including any of the following:

   * Left ventricular ejection fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
   * QTc > 480 msec on screening ECG (using the QTcF formula)
   * Angina pectoris that requires the use of anti-anginal medication
   * Ventricular arrhythmias except for benign premature ventricular contractions
   * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
   * Conduction abnormality requiring a pacemaker
   * Valvular disease with document compromise in cardiac function
   * Symptomatic pericarditis
10. Patient has a history of cardiac dysfunction including any of the following:

    * Myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    * Documented cardiomyopathy
11. Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus
12. Patient has other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol

    * Significant symptomatic deterioration of lung function. If clinically indicated, pulmonary function tests including measures of predicted lung volumes, DLco, O2 saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates.
13. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection). Patients with unresolved diarrhea will be excluded as previously indicated
14. Patient was treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
15. Patient is currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug.
16. Patients receiving chronic treatment with steroids or another immunosuppressive agent. Patients must have been off all corticosteroids (except for physiologic doses of hydrocortisone as replacement therapy) for at least 2 weeks prior to study entry.

    * Note: Single doses, or topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed.
17. Patient has taken herbal medications and certain fruits within 7 days prior to starting study drug. Herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng. Fruits include the CYP3A inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits. Regular orange juice is permitted.
18. Patient is currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug. Please refer to Table 4-8 for a list of prohibited inhibitors and inducers of CYP3A (Please note that co-treatment with weak inhibitors of CYP3A is allowed).
19. Patient received chemotherapy or targeted anticancer therapy ≤ 3 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug, and have related side effects must recover to a grade 1 or less before starting the trial
20. Patient received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) with ≤ 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy
21. Patient received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
22. Patient underwent major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy.
23. Patient is currently taking therapeutic doses of warfarin sodium or any other coumadin-derivative anticoagulant.
24. Patient is pregnant or breast feeding or is of reproductive potential and not employing an effective method of birth control.

    * Note: Double barrier contraceptives must be used through the trial by both sexes. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test ≤ 72 hours prior to initiating treatment.
    * Note: Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL [for US only: and estradiol < 20 pg/mL] or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
    * Note: Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during treatment for 4 weeks (5 T1/2) after stopping treatment. The highly effective contraception is defined as either:

      i. True abstinence: When this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

    ii. Sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.

    iii. Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate). For female subjects on the study, the vasectomised male partner should be the sole partner for that patient.

    iv. Use of a combination of any two of the following (a+b):
    1. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    2. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

       * Oral contraception, injected or implanted hormonal methods are not allowed as BKM120 potentially decreases the effectiveness of hormonal contraceptives.
25. Patient has known diagnosis of human immunodeficiency virus (HIV) infection
26. Patient has history of another malignancy within 5 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix
27. Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator
28. Patient is concurrently using other approved or investigational antineoplastic agent.
29. Patient taking or needing enzyme-inducing anti-epileptic medication.
30. Patient has an acute viral hepatitis or a history of chronic or active HBV or HCV infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-05-29 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce A. O'Shaughnessy, MD, Principal Investigator — US Oncology Research, McKesson Specialty Health; Morris D. Groves, MD, JD, Principal Investigator — US Oncology Research, McKesson Specialty Health
Locations (1):
- Please contact Zuzanne Bristow for list of sites, Multiple Locations, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- BKM120 Plus Capecitabine: BKM120 will be administered at a dose of 100 mg orally (PO) daily. Capecitabine will be administered at a dose of 1000 mg/m2 orally (PO) twice a day (rounded down to the nearest 500 mg pill) 14 days on and 7 days off.
  For patients with HER2+ MBC only, standard every 3-weekly trastuzumab (6 mg/kg IV) will be added to the capecitabine/BKM120.
  BKM120
  capecitabine
  Trastuzumab
Period: Overall Study
Arm/Group | BKM120 Plus Capecitabine
Started | 10
Completed | 4
Not Completed | 6
Not completed — Adverse Event | 3
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | BKM120 Plus Capecitabine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1
  Race: Black | 2
  Race: Caucasian | 6
  Race: Hispanic | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR)
Description: CBR in the patients following WBRT or SRS or both will be the primary endpoint and is calculated as the total number of responders (CR or PR, assessed by RECIST 1.1) plus stable disease greater than or equal to 24 weeks (CR + PR + SD ≥ 24 weeks) divided by the total number of evaluable patients.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: until disease progression (assessed by RECIST 1.1), unacceptable toxicity, death, or discontinuation from study for any other reason, up to 2 years from date of patient registration
Measure: Number (90% Confidence Interval); unit: proportion of patients with CBR
Arm/Group | BKM120 Plus Capecitabine
Number analyzed (Participants) | 10
proportion of patients with CBR | 0.1 [-0.56 to 0.256]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: To assess ORR (CR + PR) associated with BKM120 plus capecitabine in the central nervous system based on local investigator assessment. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: as for outcome 1
Measure: Number (90% Confidence Interval); unit: proportion of patients with ORR
Arm/Group | BKM120 Plus Capecitabine
Number analyzed (Participants) | 10
proportion of patients with ORR | 0.0 [0.0 to 0.0]

3. Secondary Outcome: Median Time to Progression
Description: To assess median time to progression (TTP) associated with BKM120 plus capecitabine.
Time Frame: as for outcome 1
Measure: Median (Standard Deviation); unit: months
Arm/Group | BKM120 Plus Capecitabine
Number analyzed (Participants) | 10
months | 5.59 (4.64)

4. Secondary Outcome: Median Overall Survival
Description: To determine median overall survival (OS) associated with BKM120 plus capecitabine.
Time Frame: up to 2 years from date of patient registration
Measure: Median (Standard Deviation); unit: months
Arm/Group | BKM120 Plus Capecitabine
Number analyzed (Participants) | 10
months | 11.135 (6.302)

5. Secondary Outcome: Number of Treatment-related Serious AEs
Description: To characterize the safety and tolerability of BKM120 plus capecitabine, with or without trastuzumab
Time Frame: as for outcome 1
Measure: Number; unit: Number of Treatment-related Serious AEs
Arm/Group | BKM120 Plus Capecitabine
Number analyzed (Participants) | 10
Number of Treatment-related Serious AEs | 7

ADVERSE EVENTS:
Time Frame: until 30 days after last dose of patient's study treatment, for up 2 years from date of registration (enrollment into study)
Arm/Group | BKM120 Plus Capecitabine
All-Cause Mortality (participants affected / at risk) | 7/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BKM120 Plus Capecitabine (N=10)
Colitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weakness generalized (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 2 (2)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BKM120 Plus Capecitabine (N=10)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypovolemia (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Disorder ear (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Disorder eye (Eye disorders) | 1 (1)
Eye floaters (Eye disorders) | 1 (1)
Vision abnormal (Eye disorders) | 1 (1)
Visual disturbance (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 5 (5)
Canker sore oral (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cramp abdominal (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Spasm oropharyngeal (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5)
Falling down (General disorders) | 2 (2)
Fatigue (General disorders) | 5 (5)
Hand-foot syndrome (General disorders) | 1 (1)
Legs restless (General disorders) | 1 (1)
Taste alteration (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Bilirubin increased (Investigations) | 2 (2)
Creatinine serum increased (Investigations) | 1 (1)
ALT increased (Metabolism and nutrition disorders) | 2 (2)
Amylase increased (Metabolism and nutrition disorders) | 1 (1)
AST increased (Metabolism and nutrition disorders) | 2 (2)
Dehyrdration (Metabolism and nutrition disorders) | 2 (2)
Growth accelerated (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Lipase increased (Metabolism and nutrition disorders) | 1 (1)
Potassium deficiency (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Edema cerebral (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Neuropathy (Nervous system disorders) | 1 (1)
Numbness (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Emotional lability (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Incontinence urinary (Renal and urinary disorders) | 1 (1)
Renal function abnormal (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Facial swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/82/NCT02000882/Prot_SAP_000.pdf